CLINICAL TRIAL: NCT06132425
Title: Reward Processes and Rehearsal in Exposure Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Nora Barnes-Horowitz, MA, CPhil, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#23-000236
Record Dates: First submitted 2023-11-06; First posted 2023-11-15 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Anxiety Disorders; Public Speaking Fear
Keywords: anxiety; extinction; positive affect; reward sensitivity
MeSH Terms: conditions — Anxiety Disorders; Glossophobia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Rehearsal (Experimental): After every two exposure trials, participants will complete a rehearsal exercise prompting reflection of expectancy violation and rehearsal of the inhibitory association between the conditional stimulus (i.e., speech) and the unconditional stimulus (i.e., rejection). During rehearsal, participants are prompted to identify positive emotional experiences associated with exposure trial outcomes.
  Interventions: Behavioral: Exposure; Behavioral: Rehearsal
- Neutral Rehearsal (Active Comparator): After every two exposure trials, participants will complete a rehearsal exercise prompting reflection of expectancy violation and rehearsal of the inhibitory association between the conditional stimulus (i.e., speech) and the unconditional stimulus (i.e., rejection). During rehearsal, participants are prompted to maintain a neutral, non-emotional stance and focus on overall exposure trial outcomes.
  Interventions: Behavioral: Exposure; Behavioral: Rehearsal

INTERVENTIONS:
Behavioral: Exposure — All participants complete two study visits, each consisting of 8 exposure trials for durations of 1 minute each, resulting in a total of 16 exposures. For each exposure, participants are assigned a speech topic and given 1 minute to give an unprepared speech to two study confederates.
Behavioral: Rehearsal — After every two exposures, participants will complete a rehearsal task where the participant is asked to use a positive or neutral approach to remember and recount the exposures they have just completed.

SUMMARY:
The purpose of this study is to 1) examine the importance of self-reported relief following exposure and 2) test whether positive-focused rehearsal following exposure can improve treatment outcomes for participants who endorse fear of public speaking.

Exposure therapy is an extinction-based behavioral technique, often employed in the context of cognitive behavioral therapy. It involves strategically exposing an individual to a feared stimulus in an effort to generate new non-fear associations with that stimulus. Relief refers to the positive, rewarding emotions associated with the absence of an expected aversive outcome following exposure to a feared stimulus.

In the current study, participants will engage in a series of short public speaking exposures that take place over two sessions. After every two exposures, participants will be asked to complete either a positive or neutral rehearsal exercise, consisting of recalling either positive or neutral aspects of the speech exposures. At multiple points throughout the study, participants will complete ratings of reward sensitivity, positive affect, relief, and expectancy of the aversive outcome.

The investigators will test the following: 1) the relationship of reward sensitivity and positive affect with relief following exposures, 2) the relationship between relief after exposure and learning rate (i.e., learning that the feared stimulus does not predict an aversive outcome), 3) potential differences in exposure outcomes between the positive and neutral rehearsal groups.

DETAILED DESCRIPTION:
Treatment response rates for cognitive behavioral therapy (CBT) across anxiety disorders average approximately 50% post-treatment and at follow-up. Thus, recent research has amplified efforts toward improving treatment methodology in an attempt to optimize clinical outcomes. Many efforts have targeted exposure therapy, an evidence-based behavioral technique during which a participant is strategically and repeatedly exposed to a feared stimulus in order to generate new non-fear associations with that stimulus.

Mechanisms of exposure therapy have been conceptualized using inhibitory retrieval models of extinction learning. These models, derived from Pavlovian conditioning, posit that extinction is dependent upon formation of an inhibitory association where the feared conditional stimulus (CS) no longer predicts the aversive unconditional stimulus (US). The new inhibitory CS-noUS association then competes with the original CS-US association. Research has demonstrated that greater expectation of US occurrence (US expectancy) followed by the unexpected omission of the US (i.e., expectancy violation) is associated with greater learning of the inhibitory association. Exposure therapy is a clinical proxy of extinction; in order to compete with the original association between public speaking (CS) and rejection (US), participants engage in repeated exposures to the CS without the US (no rejection) and form a new inhibitory association wherein public speaking no longer predicts rejection. Strategies to enhance this inhibitory learning process include mental rehearsal, where information from a previous exposure trial is recounted to reinforce the newly learned inhibitory association.

There is also promising evidence which suggests that reward processes may facilitate extinction learning, though studies have yet to be conducted in a clinical sample. Experimental studies have demonstrated that greater relief, a positive emotion that occurs following US omission, is associated with greater expectancy violation. This suggests that positive emotions during exposure (e.g., relief) may directly influence the extinction learning process. Reduced positive affect has been associated with decreased updating of US expectancies, leading to slower learning during extinction. In contrast, elevated positive affect has been associated with enhanced encoding, rehearsal, and retrieval processes, which may lead to faster learning during extinction and prevent return of fear (i.e., relapse). Strategies designed to enhance reward sensitivity and positive affect may therefore be an important avenue of future research to improve exposure therapy outcomes. While not yet applied during exposure, strategies aimed to increase reward sensitivity via positive-focused rehearsal have led to decreased anxiety, depression, and negative affect and increased positive affect. Recent work has shown that rehearsal without a positive focus immediately following exposure leads to reductions in anxiety. Therefore, rehearsal following exposure that specifically focuses on positive emotions to increase reward sensitivity has the potential to lead to even greater symptom improvement.

The current study seeks to examine the role of relief during extinction learning and to test whether positive-focused rehearsal exercise may be implemented to improve treatment outcomes in exposure therapy in a population of individuals who demonstrate excessive fear of public speaking. There are three main goals of the study: 1) examine the relationship of reward sensitivity and positive affect with relief following exposures, 2) examine the relationship between relief after exposure and learning rate (i.e., learning that the feared stimulus does not predict an aversive outcome), and 3) test the efficacy of a positive rehearsal exercise following exposure compared to a neutral rehearsal exercise.

Participants will engage in a series of short public speaking exposures that take place over two sessions. After every two exposures, participants will be asked to complete either a positive or neutral rehearsal exercise, consisting of recalling either positive or neutral aspects of the speech exposures. At multiple points throughout the study, participants will complete ratings of reward sensitivity, positive affect, relief, and expectancy of the aversive outcome.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Elevated score on public speaking anxiety/avoidance screening questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Positive Rehearsal | Neutral Rehearsal
Started | 44 | 44
Visit 1 | 42 | 42
Visit 2 | 38 | 40
Follow-Up | 38 | 37
Completed | 38 | 37
Not Completed | 6 | 7
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Did not follow study instructions | 0 | 2
Not completed — Lost to Follow-up | 3 | 5

BASELINE CHARACTERISTICS:
Population: We report on baseline measures for participants who at least completed Visit 1 of the study and therefore engaged in at least one session of exposure and rehearsal exercises (n=84).
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Rehearsal | Neutral Rehearsal | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.5 (4.0) | 20.0 (2.5) | 20.2 (3.3)
Sex/Gender, Customized [Number; unit: participants]
  Sex assigned at birth, female | 35 | 39 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 10 | 24
  Not Hispanic or Latino | 28 | 32 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5
  Asian | 12 | 17 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 23 | 20 | 43
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
PHQ-8 [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire (PHQ-9; Kroenke et al., 2001) is a 9-item self-report measure of depression symptoms. An 8-item version of this measure was used for the current study that excluded the suicide item (Kroenke et al., 2009). Items were rated on a four-point Likert scale (0 = not at all; 3 = nearly every day) and summed (range of scores = 0-24), where higher scores reflect greater depression symptom severity.
  units on a scale | 8.8 (5.7) | 9.2 (5.3) | 9.0 (5.5)
LSAS [Mean (Standard Deviation); unit: units on a scale] — The Liebowitz Social Anxiety Scale (LSAS; (Liebowitz, 1987) is a 24-item self-report measure of social anxiety symptoms that assesses fear of various situations and then avoidance of those same situations (resulting in a total of 48 item ratings). Items were rated on a four-point Likert scale (0 = none/never; 3 = severe) and summed (range of scores = 0-144), where higher scores reflect greater social anxiety symptom severity.
  units on a scale | 72.4 (22.3) | 73.3 (22.9) | 72.9 (22.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Public Speaking Anxiety
Description: Responses to two self-reported questions assessing public speaking anxiety and avoidance (scored from 0-8, where higher scores reflect greater public speaking anxiety and avoidance) and responses to the Personal Report of Public Speaking Anxiety (PRPSA; scored from 34-170, where higher scores reflect greater public speaking anxiety symptom severity).
Time Frame: Baseline through study completion, an average of 3 weeks.
Population: 42 participants from each group completed baseline measures. 38 participants in the positive group and 40 in the neutral group completed post-exposure measures (6 lost to follow-up, withdrew from the study, or did not follow study instructions). 38 participants in the positive group and 37 in the neutral group completed follow-up measures (3 lost to follow-up). Additionally, 2 participants in the positive group partially completed follow-up measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Rehearsal | Neutral Rehearsal
Number analyzed (Participants) | 42 | 42
units on a scale
  Baseline public speaking anxiety | 6.5 (0.8) | 6.6 (1.0)
  Baseline public speaking avoidance | 6.2 (1.4) | 6.3 (1.2)
  Baseline PRPSA | 136.1 (14.9) | 138.8 (14.1)
  Post-exposure public speaking anxiety: number analyzed (Participants) | 38 | 40
  Post-exposure public speaking anxiety | 5.4 (1.5) | 5.3 (1.7)
  Post-exposure public speaking avoidance: number analyzed (Participants) | 38 | 40
  Post-exposure public speaking avoidance | 4.8 (1.7) | 4.3 (2.0)
  Post-exposure PRPSA: number analyzed (Participants) | 38 | 40
  Post-exposure PRPSA | 123.8 (17.9) | 122.8 (19.5)
  Follow-up public speaking anxiety: number analyzed (Participants) | 38 | 37
  Follow-up public speaking anxiety | 5.3 (1.8) | 4.8 (1.9)
  Follow-up public speaking avoidance: number analyzed (Participants) | 38 | 37
  Follow-up public speaking avoidance | 4.6 (1.9) | 4.2 (2.2)
  Follow-up PRPSA: number analyzed (Participants) | 36 | 37
  Follow-up PRPSA | 122.4 (19.3) | 119.7 (18.4)

2. Secondary Outcome: Learning Rate
Description: Learning rate was calculated by using computational modeling of a prediction error formula (e.g., Rescorla & Wagner, 1972), similar to previous approaches (Barnes-Horowitz, et al., in press; Zbozinek, Perez, et al., 2022). Prior to each exposure, participants rated their expected likelihood that their feared outcome would occur on the upcoming exposure (scores ranged from 0-100). Using computational modeling, these ratings across all exposures were then input into a prediction error formula in order to derive an estimated learning rate (i.e., rate of change in expectancy ratings across exposures) for each participant. Larger, more positive learning rate values reflect greater and faster learning via faster updating of expectancy ratings across exposures.
Time Frame: Sessions 1 through 2, an average of 2 weeks.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Positive Rehearsal | Neutral Rehearsal
Number analyzed (Participants) | 42 | 42
unitless | .17 (.19) | .24 (.19)

3. Secondary Outcome: Relief Rate
Description: Relief rate was calculated by using computational modeling of a prediction error formula (e.g., Rescorla & Wagner, 1972), similar to previous approaches (Barnes-Horowitz, et al., in press; Zbozinek, Perez, et al., 2022). After each exposure, if the feared outcome did not occur, participants rated the degree of relief they felt that their feared outcome did not occur (scores ranged from 0-100). Using computational modeling, these ratings across all exposures were then input into a prediction error formula in order to derive an estimated relief rate (i.e., rate of change in relief ratings across exposures) for each participant. Larger, more positive relief rate values reflect greater and faster updating of relief ratings across exposures.
Time Frame: Sessions 1 through 2, an average of 2 weeks.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Positive Rehearsal | Neutral Rehearsal
Number analyzed (Participants) | 42 | 42
unitless | .02 (.11) | -.001 (.06)

4. Secondary Outcome: Change in Positive Affect
Description: Change in self-reported positive affect measured using a visual analog scale (scored from 1-9 where higher scores reflect greater positive affect).
Time Frame: Baseline through session 2, an average of 2 weeks.
Population: 42 participants from each group completed baseline measures. 38 participants in the positive group and 40 in the neutral group completed post-exposure measures (6 lost to follow-up, withdrew from the study, or did not follow study instructions).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Rehearsal | Neutral Rehearsal
Number analyzed (Participants) | 42 | 42
units on a scale
  Baseline | 4.9 (2.2) | 4.5 (2.0)
  Post-exposure: number analyzed (Participants) | 38 | 40
  Post-exposure | 4.2 (2.3) | 4.4 (2.1)

5. Secondary Outcome: Change in Reward Sensitivity
Description: Change in self-reported reward sensitivity using the Positive Valence System Scale (PVSS; scored from 21-189 where higher scores reflect greater reward sensitivity).
Time Frame: Baseline through session 2, an average of 2 weeks.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Rehearsal | Neutral Rehearsal
Number analyzed (Participants) | 42 | 42
units on a scale
  Baseline | 142.9 (20.5) | 145.7 (17.9)
  Post-exposure: number analyzed (Participants) | 38 | 40
  Post-exposure | 146.3 (18.5) | 148.3 (20.4)

6. Secondary Outcome: Change in Reward Sensitivity
Description: Change in self-reported reward sensitivity was assessed using the Behavioral Activation Scale (BAS). Items were rated on a four-point Likert scale (1 = strongly disagree; 4 = strongly agree) and summed (range of scores = 13-52), where higher scores reflect greater reward sensitivity.
Time Frame: Baseline through session 2, an average of 2 weeks.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Rehearsal | Neutral Rehearsal
Number analyzed (Participants) | 42 | 42
units on a scale
  Baseline | 39.6 (5.9) | 39.9 (5.5)
  Post-exposure: number analyzed (Participants) | 38 | 40
  Post-exposure | 41.2 (6.0) | 40.5 (6.1)

ADVERSE EVENTS:
Time Frame: From baseline through study completion, an average of 3 weeks.
Arm/Group | Positive Rehearsal | Neutral Rehearsal
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/25/NCT06132425/Prot_SAP_000.pdf